CLINICAL TRIAL: NCT02710695
Title: Pain in America: A Randomized Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of available time
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Nkemakolam Egekeze, Orthopaedic Research Fellow, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-026
Record Dates: First submitted 2016-03-12; First posted 2016-03-17 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Orthopaedic Related Pain (Musculoskeletal Pain)
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Control (Active Comparator): This group will receive a 10 minute discussion
  Interventions: Behavioral: Control
- Intervention (Active Comparator): This group will receive a 10 minute standardized discussion
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Control — This group will receive a standardized 10 minute discussion.
  Arms: Control
Behavioral: Intervention — This group will receive a standardized 10 minute discussion
  Arms: Intervention

SUMMARY:
Each day orthopaedic surgeons worldwide treat patients with musculoskeletal pain. But little evidence exists about orthopaedic patient understanding of the common methods of managing musculoskeletal pain. Therefore, it is our aim to determine which discussion method best improves patient comprehension of common methods of managing pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are new to a discussion about the common methods of managing musculoskeletal pain, over the age of 18, native English speakers

Exclusion Criteria:

* Patient with a previous orthopaedic surgery or musculoskeletal pain consultation, patients without the capacity to give consent, chronic narcotic users. Patients with a severe mental, visual, auditory or tactile impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
The Nkem Musculoskeletal Pain Management Comprehension Test "NMPMCT" | 15 minutes
  Validated Questionnaire

SECONDARY OUTCOMES:
Surveys | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Nkem Egekeze, MD, Principal Investigator — UMKC Department of Orthopaedic Surgery; Charles Rhoades, MD, Study Director — UMKC Department of Orthopaedic Surgery; Mark Bernhardt, MD, Study Director — UMKC Department of Orthopaedic Surgery; Karen Williams, PhD, Study Director — UMKC Department of Orthopaedic Surgery
Locations (1):
- UMKC Department of Orthopaedic Surgery, Kansas City, Missouri, United States